CLINICAL TRIAL: NCT01480102
Title: Paravertebral Block for Percutaneous Nephrolithotomy (PRONE)
Brief Title: Paravertebral Block for Percutaneous Nephrolithotomy
Acronym: PRONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Thomas Turk, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 203648
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Post Operative Pain
Keywords: Percutaneous nephrolithotomy; Paravertebral block; bupivacaine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B- No Block (Placebo Comparator): Participants randodmized to this arm will have a local anesthetic injection and pressure applied to the paravertebral space. A paravertebral injection will not be conducted.
  Interventions: Other: Group B- No block
- Group A- Paravertebral block (Active Comparator): Participants randodmized to this arm will have a local anesthetic (Bupivicaine 0.5% without epinephrine) injection and will be given a paravetebral block into the T10 paravertebral space..
  Interventions: Drug: Group A-Paravertebral block

INTERVENTIONS:
Drug: Group A-Paravertebral block — Bupivicaine 0.5% without epinephrine (100mg)20cc will be injected into the T10 paravertebral space. Active Group
  Other Names: Group A-Paravertebral block Active Group
  Arms: Group A- Paravertebral block
Other: Group B- No block — direct pressure for 5 minutes will be held at the site of the where the local anesthetic was applied to mimic the application of the block.
  Other Names: Placebo Group
  Arms: Group B- No Block

SUMMARY:
This study will compare post-operative pain levels in patients who receive paravertebral block prior to Percutaneous Nephrolithotomy (PCNL) surgery versus those who do not receive the block. We hypothesize that patients who receive the block will have lower post-operative pain scores and require less narcotics.

DETAILED DESCRIPTION:
The strategies used to manage nephrolithiasis including medical expulsive therapy, extracorporeal shock wave (ESWL), ureteroscopy, open surgery and percutaneous nephrolithotomy (PCNL). PCNL in an inpatient procedure performed in two steps. Step 1, is the placement of a drainage line (nephrostomy tube) from the back into the collecting system of the kidney. This step is typically performed by interventional radiologists under conscious sedation. Step 2 is performed by urologists and involves dilating the tract of the nephrostomy tube, placement of an access sheath and actual removal of the stone using endoscopic equipment. The minimally invasive approach of PCNL is well accepted to be as effective as open procedures for stone removal with less morbidity. Post-operative pain management remains challenging and can lead to extended hospital stays.

This randomized, double-blinded trial designed to assess the effects of paravertebral block on intra-operative and post-operative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Consent to undergo percutaneous nephrolithotomy
* Between the ages of 18 and 75
* Able to consent, fill out study documents, and complete all study procedures and follow-up visits

Exclusion Criteria:

* Will have bilateral percutaneous nephrolithotomy
* Have an infection at the site of the proposed block
* Have anatomy that prevents ability to perform block
* Have a coagulopathy which may increase their chances of bleeding from the block
* Have a known allergy to local anesthetics
* Are unable to fill out the VAS scale due to physical or mental conditions
* Are unable to use a patient controlled analgesia (PCA) device due to physical or mental conditions
* Are pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-08; Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 24 hours
  post-operative pain will be measured by the Visual Analog Scale (VAS.

SECONDARY OUTCOMES:
Opiod Use | 24 hours
  All patients will receive the same post-operative pain control, which does not deviate from our standard protocol for patients receiving PCNL. All patients will be immediately given a PCA in recovery. Patients allergic to morphine/dilaudid will be given a narcoticopioid substitute (that will be converted to morphine equivalents for the purpose of the study). Nurses will be allowed to administer IV boluses of morphine PRN for inadequate pain control. If four boluses did not yield adequate analgesia, fentayl 50mcg will be used until adequate pain control is achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turk, Principal Investigator — Loyola Medical Center
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided